CLINICAL TRIAL: NCT01484860
Title: A Phase II Single Arm Study of AUY922 in Patients With Metastatic Pancreatic Adenocarcinoma Who Are Resistant to First Line Chemotherapy
Brief Title: Study of AUY922 in Metastatic Pancreatic Cancer Who Are Resistant to First Line Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DDP-922
Record Dates: First submitted 2011-11-10; First posted 2011-12-02 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Adenocarcinoma of the Pancreas; Metastatic Disease
Keywords: AUY922; Pancreas; Pancreatic cancer; Adenocarcinoma of the pancreas; Cancer of the pancreas; Metastatic; Advanced; Advanced disease; Prior systemic anticancer therapy
MeSH Terms: conditions — Neoplasm Metastasis; Pancreatic Neoplasms | interventions — 5-(2,4-dihydroxy-5-isopropylphenyl)-4-(4-morpholin-4-ylmethylphenyl)isoxazole-3-carboxylic acid ethylamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AUY922 (Experimental): AUY922 will be administered as a weekly infusion at a dose of 70 mg/m2 based on the recommended phase II dose from the phase I study or alternate dose based on the phase I study final results.The drug will be continued until disease progression or unacceptable toxicity. One cycle will be defined as 4 weeks of treatment.
  Interventions: Drug: AUY922

INTERVENTIONS:
Drug: AUY922 — AUY922 is a solution for intravenous administration Dose: 70 mg/m2 over 1 hour, weekly

SUMMARY:
This is a phase II study to see how useful study drug AUY922 is in patients with metastatic pancreatic cancer who have received or are intolerant to first-line chemotherapy.

AUY922 is an intravenous drug that blocks a protein called heat shock protein 90 (Hsp90). Hsp90 works by keeping a number of other proteins stable and active, including many proteins that are involved in tumor growth and death. When Hsp90 is blocked from working, it is believed that many of the other proteins that it stabilizes will also be blocked, which will cause tumor growth to slow or stop.

During the study, patients will visit the clinic once a week, every 4 week cycles to receive AUY922 intravenously and to have tests and procedures done. As part of the study, archived tumor tissue will be collected and patients will be asked to have blood samples taken for pharmacokinetic testing. Patients will be invited to take part in an optional banking of blood samples for future studies.

The primary hypothesis of this study is that AUY922 improves disease control rate compared with what would be expected from best supportive care.

DETAILED DESCRIPTION:
This is a single arm open label Phase II clinical trial evaluating the efficacy of AUY922 in patients with advanced pancreatic cancer who have been previously treated with or are intolerant to first line chemotherapy. The primary objective is to assess the efficacy of this agent by assessing the disease control rate (DCR) (objective response plus prolonged stable disease (>16 weeks).

The current standard therapy for patients who have advanced, metastatic or inoperable pancreatic cancer previously treated with or intolerant to first line chemotherapy is best supportive care. New treatment options are urgently needed.

Heat shock protein 90 (HSP90) is an ATP-dependent molecular chaperone protein involved in the stabilization of a number of membrane and intracellular proteins including HER2, BCR-ABL, C-SRC, EGFR, RAF, VEGFR, AKT, and RAS. Many of these proteins are highly expressed in pancreatic adenocarcinoma.

AUY922 is a novel isoxazole-based HSP90 inhibitor. AUY922 acts by inhibiting HSP90 ATPase activity (IC50 of 30 nm) and preventing the formation of a multichaperone complex between HSP90 and other heat shock proteins. This then prevents HSP90 from performing its functions on client proteins.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of adenocarcinoma of the pancreas with metastatic disease
* Patients have received at least one prior systemic anticancer therapy for their advanced disease, which may include a gemcitabine based or 5-FU based therapeutic regimen. Patients with resected disease who relapse within 6 months of completion of adjuvant gemcitabine would also be eligible.
* Patients with progressive disease (radiological confirmation required) after at least one line of chemotherapy for pancreatic adenocarcinoma. Patients must have at least one measurable lesion as defined by RECIST criteria. Irradiated lesions are only evaluable for disease progression.
* Patient's age is ≥ 18 years of age
* Patients may have received prior radiation treatment for management of local disease providing that disease progression has been documented, all toxicities have resolved, to ≤ grade 1 and the last fraction of radiation treatment was completed at least 4 weeks prior to randomization (2 weeks for palliative radiotherapy).
* ECOG performance status of 0 or 1.
* Life expectancy of greater than 12 weeks
* Patients must have following laboratory values within 7 days prior to starting treatment:

  * Hematological:
  * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
  * Hemoglobin (Hgb) ≥ 90 g/L
  * Platelets (plt) ≥ 100 x 109/L
  * Biochemistry:
  * Potassium within normal limits
  * Total calcium (corrected for serum albumin) and Phosphorus within normal limits
  * Magnesium above LLN or correctable with supplements
  * Adequate liver function defined as:
  * AST/SGOT and ALT/SGPT ≤ 1.5 x Upper Limit of Normal (ULN)
  * AST/SGOT and ALT/SGPT ≤ 2.5 x Upper Limit of Normal (ULN) if liver metastases are present
  * Serum bilirubin ≤ 1.5 x ULN
  * eGFR ≥ 50 mL /min
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to randomization. Postmenopausal women must have been amenorrheic for ≥ 24 months in order to be considered "of non-childbearing potential". This should be documented appropriately in the patient's medical history.

Exclusion Criteria:

* Patients with a history of another primary malignancy that is clinically significant or requires active intervention
* Prior treatment with any HSP90 or HDAC inhibitor compounds, including valproic acid
* Patients with a significant history of cardiac disease, including:

  * Impaired cardiac function, including any one of the following:
  * History (or family history) of long QT syndrome
  * Mean QTc ≥ 450 msec on baseline ECG
  * History of clinically manifested ischemic heart disease ≤ 6 months prior to study start
  * History of heart failure or left ventricular (LV) dysfunction (LVEF ≤ 45%) by MUGA or ECHO
  * Clinically significant ECG abnormalities
  * History or presence of atrial fibrillation, atrial flutter or ventricular arrhythmias including ventricular tachycardia or Torsades de Pointes
  * Other clinically significant heart disease (e.g. congestive heart failure, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
  * Clinically significant resting bradycardia (< 50 beats per minute)
  * Patients who are currently receiving treatment with any medication which has a relative risk of prolonging the QTc interval or inducing Torsades de Pointes and cannot be switched to an alternative drug or discontinued prior to commencing start of treatment.
  * Obligate use of a cardiac pacemaker
* Patients with a serious active infection at the time of registration or other serious underlying medical conditions that would impair the ability of the patient to receive protocol treatment.
* Patients with a known central nervous system metastases. CT scan of the brain is NOT required unless there is suspicion of CNS metastases.
* Patients with any condition (e.g. psychological, geographical, etc.) that does not permit compliance with the protocol.
* Pregnant or lactating females.
* Women of child bearing potential or sexually active males who are not employing adequate contraception. Adequate methods of contraception include use of oral contraceptives or Depot-Provera, with an additional barrier method (diaphragm with spermicidal gel OR condoms with spermicide); a double-barrier method (diaphragm with spermicidal gel AND condoms with spermicide); partner vasectomy and total abstinence.
* Patients who received systemic anti-cancer treatment prior to the first dose of study medication within the following time frames:

  * Radiotherapy, conventional chemotherapy: within 4 weeks
  * Palliative radiotherapy: within 2 weeks
  * Monoclonal antibodies: within 4 weeks
  * Nitrosoureas and mitomycin: within 6 weeks
  * Targeted agents or investigational dugs: within 4 weeks
* Patients who have had any surgery within 2 weeks prior to registration or who have not recovered from such therapy.
* Patients known to be HIV positive. Testing is not required in the absence of clinical signs and symptoms suggestive of HIV infection.
* Treatment with therapeutic doses of coumarin-type anticoagulants. (Maximum daily dose of 2 mg, for line patency permitted)
* Patients with known disorders due to a deficiency in bilirubin glucuronidation (e.g. Gilbert's syndrome)
* Unresolved diarrhea ≥ CTCAE grade 2 within 72 hours prior to registration
* Patients with acute or chronic renal disease. Chronic renal disease will be defined as patients who have stable creatinine ≥ to 1.5 ULN and/or eGFR ≤ 50mL/min. Acute renal disease will be defined as patients that have an acute (within less then 4 weeks) rise in creatinine to ≥ 1.5 ULN and/or eGFR ≤ 50mL/min, that has not resolved to the previously normal baseline levels.
* Patients with active liver disease that requires intervention.
* Patients who cannot give informed consent (i.e. mentally incompetent patients, or those physically incapacitated such as comatose patients). Patients competent but physically unable to sign the consent form may have the document signed by their nearest relative or legal guardian. Each patient will be provided with a full explanation of the study before consent is requested.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Determine anti-tumor activity using disease control rate | 18-20 months
  Disease control rate is defined as objective response rate plus prolonged stable disease (≥16 weeks).

SECONDARY OUTCOMES:
Determine safety and tolerability of AUY922 | 18-20 months
  Number of participants with adverse events. Frequency, severity and grading of adverse events. Number of participants requiring dose reductions.
Progression Free Survival | 18-20 months
  Determine antitumor activity of AUY922 using duration of time from start of treatment to time of progression or death (progression-free survival).
Overall Survival | 18-20 months
  Determine antitumor activity of AUY922 using median time from date of enrollment to date of death (overall survival)
Stable Disease Duration | 18-20 months
  Median time from date of enrollment to date of disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm J. Moore, M.D., Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada